CLINICAL TRIAL: NCT05300464
Title: A Clinical Investigation (multicentric, Single Arm, Prospective, Stratified) to Confirm the Ability of MammoWave (microwave Mammogram) in Breast Lesions Detection
Brief Title: A Clinical Investigation to Confirm the Ability of MammoWave in Breast Lesions Detection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umbria Bioengineering Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UBT 2022-01
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinical investigation with Medical Device class IIa marked CE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): All patients perform standard breast screening and also MammoWave exam.
  Interventions: Device: Clinical investigation medical device class IIa marked CE

INTERVENTIONS:
Device: Clinical investigation medical device class IIa marked CE — Patients should perform MammoWave exam. A short visit should be performed and during this visit a qualitative differentiation would be performed between patients with high density breast, and patients with low density breast. After the patients are ready for MammoWave exam. The exam will composed of two phases: the acquisition and data processing. During the acquisition that sholud takes about 10 minutes the patients would be lying in a prone position, on a bed which is part of the MammoWave. The upper part of MammoWave has a container cup shape, which contains the breast, which also has the function of separate it from the internal parts of the device. After patient is on the bed and MammoWave would start to perform the acquisition. Once the acquisition is completed, the data will be processed through an imaging algorithm, which is integrated in the device. The final output will be composed by one or more images, plus one or more parameters describing the images.

SUMMARY:
This is a multicentric, single arm, prospective, stratified by breast density clinical investigation to confirm the ability of the microwave mammogram 'MammoWave' to detect breast lesions.

MammoWave is a innovative medical device, class IIa marked CE, which uses microwaves instead of ionazing radiation (x-ray) for breast lesions. Specifically MammoWave employs a novel technique wich generates images by processing very low power (<1mW) microwave.

The MammoWave exam takes few minutes for breast and is performed with the patient lying in a confortable facing down position.

MammoWave is safe to be used at any age, in any condition (pregnancy, specific illness and for unlimited number of times.

DETAILED DESCRIPTION:
The maximum number of participants to the clinical investigation will be 600 (for all the sites). The study will be composed of two phases: a preliminary phase to 'optimize the imaging algorithm for each apparatus installed at each centre', where 15 volunteers (in each centre) having breast with no lesions (NL) will be examined by MammoWave. In the second phase, the remaining people will be enrolled (BL will be 50% of total) and examined by MammoWave by the clinical investigator, and results will be compared with the effective diagnosis already obtained by standard clinical methods. BL includes malignant lesions (BC) and benign lesions, and may be palpable or non-palpable lesions. BL includes also isolated clustered microcalcifications.

The primary gol of the clinical study is to assess MammoWave's ability in BL detection.

The study will involve investigational sites in Italy, Germany and Spain.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent Form
* Women
* Adult ≥ 18 years old
* Having a radiologist study output obtained using mammography within the last month. Such radiologist study output may be integrated with ultrasound and /or magnetic resonance imaging output if deemed necessary by the responsible investigator and when available. The radiological output will be integrated with histological one if deemed necessary by the responsible investigator and when available.
* Patients willing to comply with study protocol and recommendations

Exclusion Criteria:

* Patients who belong to any vulnerable group
* Patients with implanted electronic devices
* Patients who have undergone biopsy less than one week before MammoWave scan
* Patients with nipple piercings (unless they are removed prior to examination)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
MammoWave sensitivity (number of 'true positive' results) | During the procedure
  MammoWave sensitivity (number of 'true positive' results) compared to Reference Standard

SECONDARY OUTCOMES:
MammoWave specificity and sensitivity | During the baseline
  MammoWave specificity and sensitivity (against Reference Standard)
Sensitivity for each breast density group | During the baseline
  Sensitivity of MammoWave according to different types of breast density groups
Sensitivity for patients which had recent mammography | During the baseline
  Sensitivity for patients which had performed recently mammography exam
Patient satisfaction questionnaire | During the baseline
  Patient satisfaction questionnaire output according to their experience performing
MammoWave sensitivity in BC | During the baseline)
  Sensitivity of MammoWave in Breast Cancer detection (against reference standard)
MammoWave specificity and sensitivity using RadioSpin simulator | During the Baseline
  Specificity and sensitivity of MammoWave (against Reference Standard) when retrospectively using MammoWave data in one RadioSpin technology simulator / Artificial Intelligence (AI) algorithms. NOTE: RadioSpin (Deep oscillatory neural networks computing and learning through the dynamics of RF neurons interconnected by RF spintronic synapses) is one of the projects funded by EU within the call FUTURE EMERGING TECHNOLOGIES (FET) H2020-FETPROACT. The RadioSpin project aims to build a hardware neural network, as a "Hardware Artificial Intelligence" will be implemented. During the project, these hardware neural networks will be optimized and tested on MammoWave data, being UBT partner of RadioSpin consortium (Grant agreement ID: 101017098)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - IRCCS Policlinico San Martino, Genova, Genova
  - Ospedale San Giovanni Battista - USL Umbria 2, Foligno, Perugia
- Hospital Universitario de Toledo, Toledo, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez Sanchez-Bayuela D, Ghavami N, Romero Castellano C, Bigotti A, Badia M, Papini L, Raspa G, Palomba G, Ghavami M, Loretoni R, Calabrese M, Tagliafico A, Tiberi G. A Multicentric, Single Arm, Prospective, Stratified Clinical Investigation to Confirm MammoWave's Ability in Breast Lesions Detection. Diagnostics (Basel). 2023 Jun 17;13(12):2100. doi: 10.3390/diagnostics13122100. PMID 37370995